CLINICAL TRIAL: NCT07362342
Title: RIght VEntricle Response to Major Lung Resection in VATS and Robotic Surgery (the RIVER-2 Study)
Brief Title: RIght VEntricle Response to Major Lung Resection in VATS and Robotic Surgery
Acronym: RIVER-2
Status: Not yet recruiting | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Fulvio Nisi, Istituto Clinico Humanitas
Other Study IDs: 4590
Record Dates: First submitted 2026-01-15; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Lung Surgery; Right Ventricular Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Major pulmonary resection is associated with high postoperative morbidity and mortality, mainly due to cardiorespiratory complications. Right ventricular (RV) function is closely related to pulmonary artery pressure and tone, and it is particularly sensitive to changes in afterload. An increase in RV flow resistance can lead to acute RV dilation and reduced left ventricular compliance, potentially progressing to cardiogenic shock. In a previous study (RIVER), it was observed that increased afterload following open thoracic surgery reduces RV function, although this impairment remains subclinical. The aim of this study is to investigate the same parameters in patients with severe cardiovascular comorbidities undergoing pulmonary resection via minimally invasive approaches (VATS and robotic surgery) compared to open thoracotomy.

DETAILED DESCRIPTION:
* Major lung resection is associated with high postoperative morbidity and mortality and significant long-term decreased functional capacity, especially due to cardiorespiratory complications [2]. An overall cardiovascular performance assessment is usually carried out before this type of surgery, along with pulmonary function tests. In such a context, close attention to the right ventricle (RV) function is recommended.
* The RV is known to be exquisitely sensitive to changes in afterload[3,4]. Since RV ejection, pulmonary artery pressure (PAP), and tone are tightly coupled, an impairment in pulmonary vascular reserve can compromise RV ejection, increasing right atrial pressure and limiting maximal cardiac output [5]. We know that during acute massive pulmonary embolism (PE), the acute increase in RV outflow resistance causes acute RV dilatation and, using ventricular interdependence, markedly decreased left ventricle (LV) compliance, rapidly spiraling to acute cardiogenic shock and death. We want to explore if during major lung surgery such maneuvers as pulmonary artery branch clamping could bring to the same event. Furthermore, a postoperative RV disfunction (RVD) has been observed after open major lung surgery; in our previous study we showed that the observed increase in afterload reduced the post-operative RV function after open surgery (thoracotomy), but the impairment remained subclinical, with the RV failure being rarely observed[3].
* More in general, this effect has been investigated in literature and all studies agree with the conclusion that the postoperative RV disfunction is common after major lung surgery but there is no evidence of acute cardiogenic shock[4-9], neither during clamping nor in the port-operative period, suggesting that the mechanisms involved in the RV response are various (not just RV resistances) and, to date, not well defined. Little is known on RV disfunction after video-assisted thoracoscopic surgery[10].
* With this study our aim is to observe the difference in RV disfunction after mini-invasive video-assisted thoracic surgery (VATS and robotic surgery) compared to the open surgical approach, in the hypothesis that the thoracic compliance plays an important role in the cardio-pulmonary balance and it could be more impaired during open surgery.

RATIONALE To understand whether and to what extent RV dysfunction occurs after surgery in patients undergoing mini-invasive thoracic surgery and to compare RV function alterations after mini-invasive thoracic surgery to the open apporach.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years
* Scheduled for elective lobectomy (or bilobectomy) via minimally invasive or open thoracic surgery
* Ability to provide written informed consent at the time of hospital admission
* Moderate to high cardiopulmonary risk, defined by at least one of the following criteria:

  * ASA physical status classification 3
  * Predicted postoperative FEV1 <60% and 6-minute walk test <400 m or cardiopulmonary exercise test <20 ml/kg/min
  * DASI index <34
  * RCRI >2
  * Coronary artery disease
  * Heart failure
  * Right ventricular systolic dysfunction (TAPSE <17 mm and/or S' wave on TDI <10 cm/s)
  * Left ventricular systolic dysfunction (EF <55%)

Exclusion Criteria

* Urgent/emergency surgery
* History of pulmonary embolism
* Previous right or left pneumonectomy
* Previous lobectomy
* Completion pneumonectomy
* Pregnancy (confirmed or suspected)
* History of severe pulmonary hypertension (PAPs >40 mmHg)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective observational study in patients undergoing elective major thoracic surgery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Echocardiographic Measurement of RV dysfunction | 1 year
  Measurement of TAPSE and/or S' wave using Tissue Doppler Imaging (TDI); TAPSE/PAPs ratio